CLINICAL TRIAL: NCT04056520
Title: Clinical and Radiological Outcomes of Posterior Cervical Fusion with Medtronic Infinity Occipitocervical-Upper Thoracic (OCT) System
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Andrew Grossbach, Principal Investigator / Assistant Clinical Professor, Ohio State University
Other Study IDs: 2019H0161
Record Dates: First submitted 2019-07-23; First posted 2019-08-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Arm 1: Subjects undergoing posterior cervicothoracic fusions between C2 and upper thoracic will be enrolled
  Interventions: Device: Medtronic Infinity Occipitocervical-Upper Thoracic System using the O-arm Imaging System and StealthStation Navigation system

INTERVENTIONS:
Device: Medtronic Infinity Occipitocervical-Upper Thoracic System using the O-arm Imaging System and StealthStation Navigation system — The INFINITY™ OCT System is intended to provide immobilization and stabilization of spinal segments as an adjunct to fusion for the following acute and chronic instabilities of the craniocervical junction, the cervical spine (C1 to C7), and the thoracic spine from T1-T3:
  * Traumatic spinal fractures and/or traumatic dislocations.
  * Instability or deformity.
  * Failed previous fusions (e.g. pseudarthrosis).
  * Tumors involving the cervical spine.
  * Degenerative disease, including intractable radiculopathy and/or myelopathy, neck and/ or arm pain of discogenic origin as confirmed by radiographic studies, and degenerative disease of the facets with instability.

SUMMARY:
This study is being done to prospectively collect data on subjects having posterior cervical fusion surgery using the Medtronic Infinity system. Researchers plan to collect information from patients having this type of surgery in order to learn more about patient how patients do after the surgery, including the rate of bone healing following surgery.

The goal is for 250 patients to take part in the study or for 500 screws to be used, whichever comes first. Each patient will need a varying amount of screws to be used during their surgery. Because we are measuring the accuracy of each individual screw and the surgeon will likely use multiple screws during each surgery, it is likely that the study will reach its goal of 500 screws before 250 patients are enrolled in the study.

DETAILED DESCRIPTION:
This is a prospective single arm study of clinical and radiological outcomes as well as surgical data from posterior cervical fusion for treating degenerative disc disease (DDD). Patients undergoing posterior cervicothoracic fusions between C2 and upper thoracic will be enrolled.

Patients will be enrolled up to 250 patients (at maximum) or 500 screws, whichever is achieved first. This will adequately power the study assuming 95% screw accuracy, which is in line with published data, and assuming precision of +/- 2% with a confidence level of 9%.

The primary objective of this study is to show that the Medtronic Infinity System is safe and effective in posterior cervicothoracic fusion surgeries. Outcomes measures and complication rates will be compared to historical controls. Secondary objectives include screw accuracy rates/revision rates which can also be compared to historical controls. Other secondary objectives aim to clarify the workflow and operative time of using the O-arm and Stealth navigation for these types of cases.

Subjects will be monitored for adverse events throughout the duration of the study, particularly at and around the time of standard of care clinical assessments. The number of CT related adverse events will be evaluated. The monitoring will be performed by the investigator and study clinical research coordinator. The monitoring will occur both when a quarter and a half of the study patients have been enrolled. The study will be stopped should any significant CT related adverse events be identified.

The following data will be collected

Patient demographic and pre-operative clinical information will include:

* Name
* Age
* Sex
* Race (self-reported)
* Vitals
* Height, weight and body mass index (BMI)
* General medical/surgical history
* Medication regimen
* Smoking status (current, former, never)
* History of alcohol/substance abuse
* PROMIS
* Neurological Assessment (strength, sensory, reflexes, Hoffmann's response, Spurling's test)
* Duration of disease
* X-rays, CT, and MRI as available

Patient surgical details to be collected will include:

* Diagnosis
* Date of surgery
* Operative Index levels
* Operative time (incision open to close)
* Implants used
* Length of hospital stay
* Estimated blood loss / Surgical complications
* Somatosensory and motor intraoperative monitoring reports

Post-operative clinical information will include:

* Medication regimen
* PROMIS
* Neurological Assessment (strength, sensory, reflexes, Hoffmann's response, Spurling's test)
* X-rays, CT, and MRI as available

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Symptomatic multi-level degenerative spondylosis necessitating posterior cervical arthrodesis in the subaxial cervicothoracic spine (between C2-upper thoracic).
* Surgery performed within the Department of Neurological Surgery at The Ohio State University Wexner Medical Center (OSUWMC)

Exclusion Criteria:

* Traumatic injury
* Co-morbidity requiring medication use that may interfere with bone or soft tissue healing (i.e., high dose oral or parenteral glucocorticoids, immunosuppressive agents, methotrexate) - at discretion of investigator
* Severe co-morbidities (e.g., heart, respiratory, or renal disease)
* Clinically diagnosed osteoporosis
* Recent (<3 yrs) or co-incident spinal tumor or infection
* Concurrent involvement in another investigational drug or device study that could confound study data
* History of substance abuse (recreational drugs, prescription drugs or alcohol) that could interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up
* Subjects who are pregnant or plan to become pregnant in the next 24 months
* Prisoner
* Other contraindications for Medtronic Infinity System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing posterior cervicothoracic fusions between C2 and upper thoracic will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Related Adverse Events | 49 Days
  All Procedure related adverse events
Upper and Lower Extremity Motor Exam | 49 Days
  MMT Score 1-5 where higher score represents better outcome
Sensory Function | 49 Days
  Sensory Function Score 0-2 where higher score represents better outcome
Reflexes Score | 49 Days
  Reflex Score 0-4 where a score of 2 represents best outcome
PROMIS - 29 Profile v2.0 Physical Functioning Subscore | 49 Days
  Disease non-specific measure of health related physical functioning presented as T-scores with a mean of 50 and standard deviation of 10 with a higher score indicating better outcome
PROMIS - 29 Profile v2.0 Ability to Participate Subscore | 49 Days
  Disease non-specific measure of health related ability to participate presented as T-scores with a mean of 50 and standard deviation of 10 with a higher score indicating better outcome
PROMIS - 29 Profile v2.0 Anxiety Subscore | 49 Days
  Disease non-specific measure of health related anxiety presented as T-scores with a mean of 50 and standard deviation of 10 with a lower score indicating better outcome
PROMIS - 29 Profile v2.0 Depression Subscore | 49 Days
  Disease non-specific measure of health related depression presented as T-scores with a mean of 50 and standard deviation of 10 with a lower score indicating better outcome
PROMIS - 29 Profile v2.0 Fatigue Subscore | 49 Days
  Disease non-specific measure of health related fatigue presented as T-scores with a mean of 50 and standard deviation of 10 with a lower score indicating better outcome
PROMIS - 29 Profile v2.0 Sleep Subscore | 49 Days
  Disease non-specific measure of health related sleep presented as T-scores with a mean of 50 and standard deviation of 10 with a higher score indicating better outcome
PROMIS - 29 Profile v2.0 Pain Intensity Subscore | 49 Days
  Disease non-specific measure of health related pain intensity presented as T-scores with a mean of 50 and standard deviation of 10 with a lower score indicating better outcome
Cervical Sagittal Alignment | 49 Days
  Cervical Sagittal Alignment measured on pre- and post-operative radiographs
Hoffmann's Response Test | 49 Days
  Hoffmann's Response Test measured as Positive or Negative with negative representing the better outcome
Spurling's Compression Test | 49 Days
  Spurling's Compression Test measured a Positive or Negative with negative representing the better outcome
All Adverse Events | 49 Days
  All Adverse Events and Serious Adverse Events for study duration

SECONDARY OUTCOMES:
Modified Gerzbein & Robbins Scale | 49 Days
  Screw placement accuracy assessed using modified Gertzbein & Robbins Scale with a score range of 0-4 with lower score indicating better outcome
Screw Placement Time | 49 Days
  Time to place screw
Screw Intra-op Repositioning Rate | 49 Days
  Rate of Screw Repositioning Intraoperatively
Reference Frame Setup (Level of positioning) | 49 Days
  Level of Surgical Positioning
Perioperative AEs | 30 Days
  Rate of Perioperative AEs within 30 days post-op
OR Time | 30 Days
  Time from surgical procedure start to end
Blood Loss | 30 Days
  Blood Loss during surgery measured in cc
Length of Stay | 30 Days
  Length of Hospital Stay measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Grossbach, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waschke A, Walter J, Duenisch P, Reichart R, Kalff R, Ewald C. CT-navigation versus fluoroscopy-guided placement of pedicle screws at the thoracolumbar spine: single center experience of 4,500 screws. Eur Spine J. 2013 Mar;22(3):654-60. doi: 10.1007/s00586-012-2509-3. Epub 2012 Sep 23. PMID 23001415
- [Background] Silbermann J, Riese F, Allam Y, Reichert T, Koeppert H, Gutberlet M. Computer tomography assessment of pedicle screw placement in lumbar and sacral spine: comparison between free-hand and O-arm based navigation techniques. Eur Spine J. 2011 Jun;20(6):875-81. doi: 10.1007/s00586-010-1683-4. Epub 2011 Jan 21. PMID 21253780
- [Background] Luther N, Iorgulescu JB, Geannette C, Gebhard H, Saleh T, Tsiouris AJ, Hartl R. Comparison of navigated versus non-navigated pedicle screw placement in 260 patients and 1434 screws: screw accuracy, screw size, and the complexity of surgery. J Spinal Disord Tech. 2015 Jun;28(5):E298-303. doi: 10.1097/BSD.0b013e31828af33e. PMID 23511642
- [Background] Gertzbein SD, Robbins SE. Accuracy of pedicular screw placement in vivo. Spine (Phila Pa 1976). 1990 Jan;15(1):11-4. doi: 10.1097/00007632-199001000-00004. PMID 2326693